CLINICAL TRIAL: NCT05236530
Title: A Phase I, Open-label, Fixed-sequence, Two-period, Crossover, Drug-drug Interaction Study to Evaluate the Effect of Multiple Doses of Ganaplacide and Lumefantrine Combination on the Pharmacokinetics of Midazolam, Repaglinide, Dextromethorphan, Metformin, Rosuvastatin and Dolutegravir in Healthy Participants
Brief Title: Drug-drug Interaction Study of Ganaplacide and Lumefantrine With Midazolam, Repaglinide, Dextromethorphan, Metformin, Rosuvastatin and Dolutegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CKAF156A2104
Record Dates: First submitted 2022-02-04; First posted 2022-02-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Malaria
Keywords: Drug-drug interaction; DDI; probe; cocktail; ganaplacide; lumefantrine; midazolam; repaglinide; dextromethorphan; rosuvastatin; metformin; dolutegravir; CYP2C8; CYP2D6; CYP3A4; OATP1B1; MATE1; Pharmacokinetic; PK; safety and tolerability; healthy participants
MeSH Terms: conditions — Malaria | interventions — Midazolam; repaglinide; Dextromethorphan; Metformin; ganaplacide; Lumefantrine; Rosuvastatin Calcium; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Each participant will receive a single oral dose of the 4-probe substrate cocktail consisting of midazolam, repaglinide, dextromethorphan and metformin in the morning of Day 1 of Period 1. In Period 2, participants will receive ganaplacide and lumefantrine combination orally once daily (q.d.) in the morning on Days 1 through 3, with a single oral dose of the 4-probe substrate cocktail co-administered on Day 3.
  Interventions: Drug: Midazolam; Drug: Repaglinide; Drug: Dextromethorphan; Drug: Metformin; Drug: Ganaplacide; Combination Product: Lumefantrine
- Cohort 2 (Experimental): Each participant will receive a single oral dose of the 2 probe substrate cocktail consisting of rosuvastatin and dolutegravir in the morning on Day 1 of Period 1. In Period 2, participants will receive ganaplacide and lumefantrine combination orally q.d. in the morning on Days 1 through 3, with a single oral dose of the 2 probe substrate cocktail co-administered on Day 3.
  Interventions: Drug: Rosuvastatin; Drug: Dolutegravir; Drug: Ganaplacide; Combination Product: Lumefantrine

INTERVENTIONS:
Drug: Midazolam — Midazolam 2 mg (1 mL of 2 mg/mL oral solution) administered as a single dose in a 4-probe cocktail in the morning in Period 1 on Day 1 and in Period 2 on Day 3.
  Arms: Cohort 1
Drug: Repaglinide — Repaglinide 0.5 mg (1 x 0.5 mg tablet) administered as a single dose in a 4-probe cocktail in the morning in Period 1 on Day 1 and in Period 2 on Day 3.
  Arms: Cohort 1
Drug: Dextromethorphan — Dextromethorphan 15 mg (10 mL of 7.5 mg/5 mL syrup) administered as a single dose in a 4-probe cocktail in the morning in Period 1 on Day 1 and in Period 2 on Day 3.
  Arms: Cohort 1
Drug: Metformin — Metformin 500 mg (1 x 500 mg tablet) administered as a single dose in a 4-probe cocktail in the morning in Period 1 on Day 1 and in Period 2 on Day 3.
  Arms: Cohort 1
Drug: Ganaplacide — Ganaplacide 400 mg (4 x 100 mg tablets) administered q.d. in Period 2 on Days 1 - 3, with the 4-probe cocktail co administered on the morning of Day 3.
  Other Names: KAF156
  Arms: Cohort 1
Combination Product: Lumefantrine — Lumefantrine 960 mg (4 x 240 mg sachets) administered q.d. on Days 1 - 3, with the 4-probe cocktail (as a single dose) co administered on the morning of Day 3.
  Other Names: LUM566
  Arms: Cohort 1
Drug: Rosuvastatin — Rosuvastatin 5 mg (1 x 5 mg tablet) administered as a single dose in a 2-probe cocktail in the morning in Period 1 on Day 1 and in Period 2 on Day 3.
  Arms: Cohort 2
Drug: Dolutegravir — Dolutegravir 50 mg (1 x 50 mg tablet) administered as a single dose in a 2-probe cocktail in the morning in Period 1 on Day 1 and in Period 2 on Day 3.
  Arms: Cohort 2
Drug: Ganaplacide — Ganaplacide 400 mg (4 x 100 mg tablets) administered q.d. in Period 2 on Days 1 - 3, with the 2-probe cocktail co administered on the morning of Day 3.
  Other Names: KAF156
  Arms: Cohort 2
Combination Product: Lumefantrine — Lumefantrine 960 mg (4 x 240 mg sachets) administered q.d. on Days 1 - 3, with the 4-probe cocktail (as a single dose) co administered on the morning of Day 3.
  Other Names: LUM566
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of ganaplacide and lumefantrine combination on the substrates of cytochrome P450 (CYP) 3A4 (midazolam), CYP2C8 (repaglinide), CYP2D6 (dextromethorphan), organic cation transporter (OCT) 1, multidrug and toxin extrusion (MATE) 1 (metformin) in Cohort 1 and a substrate of the organic anion transporting polypeptide (OATP) 1B1, OATP1B3 and Breast Cancer Resistance Protein (BCRP) transporter (rosuvastatin) and an antiretroviral drug (dolutegravir) in Cohort 2.

Results from this study will provide guidance on prescribing ganaplacide and lumefantrine combination when co-administered with substrates of the CYP enzymes (CYP3A4, CYP2C8 and CYP2D6) and transporters (OCT1, MATE1, OATP1B1, OATP1B3, and BCRP), and dolutegravir.

DETAILED DESCRIPTION:
This is an open-label, 2-cohort, fixed-sequence, 2-period, crossover, drug-drug interaction (DDI) study to evaluate the effect of multiple doses of ganaplacide and lumefantrine combination on the single-dose PK of CYP substrates (midazolam [CYP3A4 substrate], repaglinide [CYP2C8 substrate], dextromethorphan [CYP2D6 substrate]), transporter substrates (metformin [OCT1 and MATE1 substrate] and rosuvastatin [OATP1B1, OATP1B3 and BCRP substrate]) and a human immunodeficiency virus (HIV) integrase inhibitor (dolutegravir) in healthy participants.

For each cohort, the study will consist of a screening period of up to 28 days, Baseline evaluations (on Day -1 of Period 1) and 2 treatment periods which are separated by a washout period. Participants who meet the eligibility criteria at Screening will be admitted to the study site for Baseline evaluations on Day -1 of Period 1. Baseline safety assessments will be performed prior to first dosing of study treatment in Period 1.

Participants will be enrolled in 1 of 2 cohorts only. Cohort 1 Participants enrolled will receive a single oral dose of the 4-probe substrate cocktail consisting of midazolam, repaglinide, dextromethorphan and metformin on Day 1 of Period 1. There will be a washout period of at least 2 days, beginning from the last PK sample collection in Period 1 and continuing until the first dose of study treatment in Period 2. In Period 2, participants will receive ganaplacide and lumefantrine combination orally once daily (q.d.) on Days 1 through 3, with a single oral dose of the 4-probe substrate cocktail co-administered on Day 3. There will be 72 hours of sequential blood sampling for PK assessment of substrates starting after the 4-probe cocktail dosing in each treatment period. Blood samples for ganaplacide, its metabolites and lumefantrine PK will also be collected on Days 1 through 6 of Period 2.

All study treatments will be administered after at least 10 hours of overnight fasting and will be followed by at least 4 hours of post dose fasting.

Cohort 2 Participants enrolled will receive a single oral dose of the 2-probe substrate cocktail consisting of rosuvastatin and dolutegravir on Day 1 of Period 1. There will be a washout period of at least 2 days, beginning from the last PK sample collection in Period 1 and continuing until the first dose of study treatment in Period 2. In Period 2, participants will receive ganaplacide and lumefantrine combination orally q.d. on Days 1 through 3, with a single oral dose of the 2-probe substrate cocktail co-administered on Day 3. There will be 168 hours of sequential blood sampling for PK assessment of substrates starting after the 2-probe cocktail dosing in each treatment period. Blood samples for ganaplacide, its metabolites and lumefantrine PK will also be collected on Days 1 through 10 of Period 2.

All study treatments will be administered after at least 10 hours of overnight fasting and will be followed by at least 4 hours of post dose fasting.

Both Cohorts Safety assessments (including physical examinations, electrocardiograms (ECGs), vital signs, clinical laboratory evaluations [hematology, chemistry, coagulation and urinalysis], pulse oximetry [Cohort 1 only], blood glucose monitoring [Cohort 1 only] and adverse event [AE] and serious adverse event [SAE] monitoring) will be performed during the study.

The Study Completion evaluations will occur on Day 6 of Period 2 for Cohort 1 and on Day 10 of Period 2 for Cohort 2, followed by a post-study safety contact (e.g. follow-up telephone call, email) approximately 30 days after the last dose of study treatment. In the case of early termination, Study Completion evaluations will be conducted prior to discharge from the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Healthy male and non-childbearing potential female participants 18 to 55 years of age inclusive, at Screening.
* In good health as determined by medical history, physical examination, vital signs, ECG and clinical laboratory tests at Screening.
* Must weigh at least 50 kg with a body mass index (BMI) within the range of 18.0 to 29.9 kg/m2 inclusive, at Screening.

Key Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives or 30 days prior to first dosing of study treatment, whichever is longer.
* Known family history or presence of long QT syndrome.
* Known history or current clinically significant arrhythmias.
* History or presence of malignancy of any organ system (other than treated localized basal cell or squamous cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within 5 years of Screening, regardless of whether there is evidence of local recurrence or metastases.
* History or presence of duodenal ulcer, ulcerative colitis or Crohn's disease.
* Presence of active or uncontrolled thyroid disease.
* Has had cholecystectomy (gallbladder removed). Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Apparent total body clearance of drug from plasma following extravascular administration (CL/F) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL/F will be listed and summarized using descriptive statistics.
Apparent volume of distribution during terminal elimination phase following extravascular administration (Vz/F) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz/F will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for midazolam, repaglinide, dextromethorphan and metformin | 0 (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T^1/2 will be listed and summarized using descriptive statistics.
Observed maximum plasma concentration (Cmax) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Apparent total body clearance of drug from plasma following extravascular administration (CL/F) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL/F will be listed and summarized using descriptive statistics.
Apparent volume of distribution during terminal elimination phase following extravascular administration (Vz/F) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz/F will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for rosuvastatin and dolutegravir | 0 (pre dose) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T^1/2 will be listed and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No